CLINICAL TRIAL: NCT04502706
Title: A Phase 1 Study of GS-0189 (Formerly FSI-189) as Monotherapy and in Combination With Rituximab in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: Study of GS-0189 (Formerly FSI-189) as Monotherapy and in Combination With Rituximab in Participants With Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision to discontinue development of this molecule
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRP001
Record Dates: First submitted 2020-07-16; First posted 2020-08-06 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-05

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- GS-0189 (Monotherapy Dose Escalation, MDE) (Experimental): Relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL) participants will receive GS-0189 doses of 10, 30, or 100 mg every 2 weeks.
  Interventions: Drug: GS-0189
- GS-0189 + Rituximab (Combination Dose Escalation, CDE) (Experimental): R/R NHL participants will receive GS-0189 doses of 100, 300, 1000, 2000, and 3000 mg in combination with rituximab at 375 mg/m^2.
  Interventions: Drug: GS-0189; Drug: Rituximab
- GS-0189 + Rituximab (Pharmacokinetic (PK) Evaluation) (Experimental): R/R NHL participants will receive GS-0189 dose of up to 30 mg followed by the highest designated safe dose from the Combination Dose Escalation cohort (CDE) in combination with rituximab at 375 mg/m^2.
  Interventions: Drug: GS-0189; Drug: Rituximab
- GS-0189 + Rituximab (Alternate Schedule Evaluation, ASE) (Experimental): R/R NHL participants will receive GS-0189 every 4 weeks in combination with rituximab 375 mg/m^2. The GS-0189 dose will be determined based on the totality of safety, PK, and pharmacodynamic (PD) data from the preceding cohorts.
  Interventions: Drug: GS-0189; Drug: Rituximab
- GS-0189 + Rituximab (DLBCL Expansion) (Experimental): Diffuse large B-cell lymphoma (DLBCL) participants will receive GS-0189 in combination with rituximab 375 mg/m^2. The GS-0189 dose will be determined based on the totality of safety, PK, and PD data from the preceding cohorts.
  Interventions: Drug: GS-0189; Drug: Rituximab

INTERVENTIONS:
Drug: GS-0189 — GS-0189 will be administered intravenously.
  Other Names: FSI-189
Drug: Rituximab — Rituximab will be administered intravenously.
  Arms: GS-0189 + Rituximab (Alternate Schedule Evaluation, ASE); GS-0189 + Rituximab (Combination Dose Escalation, CDE); GS-0189 + Rituximab (DLBCL Expansion); GS-0189 + Rituximab (Pharmacokinetic (PK) Evaluation)

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of GS-0189 (formerly FSI-189) as monotherapy and in combination with rituximab in participants with relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
The study will consist of 5 parts: 1) an initial Monotherapy Dose Escalation (MDE) part, 2) a Combination Dose Escalation (CDE) part, 3) a Pharmacokinetic (PK) Evaluation part, 4) an Alternate Schedule Evaluation (ASE) part and 5) a diffuse large B-cell lymphoma (DLBCL) Expansion part.

ELIGIBILITY:
Key Inclusion Criteria:

* DLBCL, follicular lymphoma (FL), mantle cell lymphoma (MCL), or marginal zone lymphoma (MZL) relapsed/refractory (R/R) to at least 2 prior lines of therapy. Prior autologous hematopoietic cell transplantation and individuals with transformed lymphomas are permitted. Individuals must be at least 3 months out from prior autologous hematopoietic cell transplantation. Individuals with indolent lymphomas must be candidates for systemic treatment in the judgment of the treating physician.
* In the DLBCL Expansion part: DLBCL that is relapsed or refractory to at least 2 prior lines of therapy. Prior autologous hematopoietic cell transplantation and individuals with transformed lymphomas are permitted.
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2.
* For the DLBCL expansion cohort, disease must be measurable for response per Lugano criteria. For all other cohorts, disease must be measurable or assessable for response per Lugano criteria.
* Exhibit acceptable hematopoietic, liver, renal, and coagulation function as assessed by laboratory tests.

Key Exclusion Criteria:

* Individuals with active brain metastases (Individuals with stable treated central nervous system (CNS) lesions who are off corticosteroid therapy for at least 3 weeks are not considered active.
* Individuals with Burkitt's lymphoma.
* Prior treatment with a chimeric antigen receptor (CAR) T-cell therapy ≤ 90 days from first dose of study drug.
* Prior allogeneic stem cell transplant.
* Previous anticancer therapy including chemotherapy, hormonal therapy, and investigational agents within 3 weeks or at least 4 half-lives (up to a maximum of 4 weeks), whichever is longer, prior to first dose of study drug.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus.
* Prior treatment with CD47 or signal regulatory protein alpha (SIRPα)-targeting agents.
* Hypersensitivity to the active substance, to murine proteins, or to any of the other excipients of rituximab
* Significant medical diseases or conditions, as assessed by the Investigator and Sponsor, that would substantially increase the risk:benefit ratio of participating in the study.
* Rituximab-containing cohorts only: Receipt of live/attenuated vaccines within 30 days of rituximab dosing
* Has persisting toxicity related to prior therapy of Grade > 1 in severity per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Treatment-Emergent Adverse Events | Up to 11 months
  Adverse events as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Laboratory Abnormalities | Up to 11 months
Pharmacokinetic (PK) Parameter: AUClast of GS-0189 | Up to 11 months
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
PK Parameter: AUCtau of GS-0189 | Up to 11 months
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
PK Parameter: Cmax of GS-0189 | Up to 11 months
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Accumulation Ratio (AR) of GS-0189 | Up to 11 months
  AR is defined as ratio based on Cmax and AUCtau after first dose and after multiple doses.
PK Parameter: Tmax of GS-0189 | Up to 11 months
  Tmax is defined as the time (observed time point) of Cmax.
PK Parameter: AUC0-tau/D Dose-normalized AUCtau of GS-0189 | Up to 11 months
  AUC0-tau/D is defined dose normalized area under the concentration-time curve from time zero (pre dose time point of the infusion) to the end of the dosing interval.
Percentage of Signal Regulatory Protein Alpha (SIRPα) Receptor Occupancy in the Blood | Up to 11 months
Serum Concentration of GS-0189 | Up to 11 months
Rate of Anti-GS-0189 Antibody Positivity | Up to 11 months
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) as assessed by Lugano Classification response criteria for lymphomas.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of disease progression.
Progression-free Survival (PFS) | Up to 2 years
  PFS is defined as the interval from the first dose date of drug to the earlier of the first documentation of definitive disease progression or death from any cause.
Overall Survival (OS) | Up to 2 years
  OS is defined as the interval from the first dose date of drug to death from any cause.
Time to Progression (TTP) | Up to 2 years
  TTP is defined as the interval from the first dose date of drug to the earlier of the first documentation of definitive disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=SRP001